CLINICAL TRIAL: NCT07129941
Title: Transdiagnostic Group Treatment of Emotional Disorders: A Cross-sectional and Naturalistic Study of Outcome, Change Processes, and Clinical Training
Brief Title: Unified Protocol Group Treatment in a University Outpatient Clinic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REK-ID 840156
Record Dates: First submitted 2025-05-22; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-05

CONDITIONS: Emotional Disorders; Anxiety; Depression - Major Depressive Disorder
Keywords: Unified Protocol; Transdiagnostic treatment; Emotional disorders; Anxiety; Depression; Group therapy
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This is a single-arm uncontrolled naturalistic trial. All eligible patients will receive the Unified Protocol (UP) intervention, but will be randomly assigned to receive treatment from either experienced psychologists or psychology students.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unified Protocol group treatment (Experimental): The Unified Protocol (UP) is a time-limited modular treatment addressing core emotion regulation difficulties in patients with emotional disorders. There will be 8-10 patients and two or three therapists in the group. Treatment consists of one individual session of diagnostic assessment, and one or two individual preparation sessions (case formulation and goal setting), and 12 weekly 2 ½ hour group treatment sessions.
  Interventions: Behavioral: Unified Protocol

INTERVENTIONS:
Behavioral: Unified Protocol — The Unified Protocol is a transdiagnostic intervention for emotional disorders here delivered in a group format

SUMMARY:
This clinical trial aims to evaluate the effectiveness and underlying processes of change of the Unified Protocol (UP) for treating emotional disorders in a university outpatient clinic. The study will involve 140 patients receiving UP treatment in a group format, delivered either by experienced or novice therapists, along with a non-clinical control group of 45 participants. Participants will self-refer on the basis of advertisement about the study through flyers, posters, project website, social media or local news media. Outcomes will be assessed through self-report measures of well-being, symptoms, emotion regulation, and the non-specific factors of treatment credibility and therapeutic alliance. Additionally, psychophysiological measures of heart rate variability and interoception will be used to explore processes influencing treatment response. Qualitative interviews will complement the quantitative data by capturing participants' perspectives on the treatment and experiences of what contributed to change.

DETAILED DESCRIPTION:
Background Anxiety and depression are the most common mental disorders, incurring vast personal and societal costs. While effective evidence-based treatments exist, healthcare systems struggle to meet the growing demand for services. A key challenge in delivering care is that most treatments are diagnosis specific. This complicates training and implementation due to clinicians having to learn multiple treatment manuals. In addition, these single-disorder treatments may also often have poor applicability to the complex symptoms and patterns of comorbidity typically seen in real-world clinical settings. As a response to these challenges, several transdiagnostic treatment protocols have been developed to target psychological processes underlying different diagnoses. One such model is the "Unified Protocol for Transdiagnostic Treatment of Emotional Disorders" (UP) developed by David Barlow and colleagues. UP addresses the functional processes that maintain emotional disorders, such as negative reactions to emotions and avoidance behaviors.

The Unified Protocol (UP) has shown non-inferiority to diagnosis-specific CBT and superiority to treatment as usual in both individual and group formats. Meta-analyses confirm its effectiveness for comorbid emotional disorders and suggest potential for cost-effective, scalable implementation.

Knowledge gaps

* Norwegian Setting: Only one small feasibility study of UP has been conducted in Norway. A larger naturalistic trial is needed to assess outcomes (quality of life, functioning, symptoms) and potential negative effects in a public health context.
* Processes of Change: More research is needed to identify active treatment mechanisms (e.g., emotion regulation, mindfulness, cognitive flexibility) and their association with outcomes in group UP. Non-specific factors such as credibility and group alliance also require investigation.
* Psychophysiological Measures: UP's impact on objective emotion regulation markers (e.g., heart rate variability, interoception) is unexplored. Inclusion of such measures can reduce bias and clarify underlying mechanisms.
* Novice Therapists: The ability of graduate psychology students to deliver UP with high fidelity in group format remains unclear and merits further investigation.

Study objectives This study aims to explore outcomes, processes of change, and user experiences of UP group treatment for patients with emotional disorders in a naturalistic clinical sample in a Norwegian setting. Additionally, it will compare the clinical sample to a healthy control group to better understand how transdiagnostic characteristics serve as vulnerability or resilience factors in the development of emotional disorders. Lastly, the study examines whether novice therapists can be trained to deliver the treatment with high levels of fidelity based on ratings of adherence and competence.

Main aims and research questions i. Assessing treatment effectiveness: To determine whether UP group treatment leads to improvements in key clinical outcomes, identify factors that influence these outcomes, and assess any negative treatment effects.

Research questions:

* Does UP group treatment lead to improvements in quality of life, everyday functioning, emotion regulation, and self-reported symptoms?
* To what extent do clinical and demographic factors impact treatment adherence and outcome?
* What type and frequency of negative treatment effects do participants report?

ii. Examining processes of change: To investigate the role of emotion regulation, interoception, and UP skill use as predictors and mediators of treatment outcomes, using both self-report and objective measures.

Research questions:

* Specific factors: To what extent do changes in UP-relevant skills and processes (e.g., emotion regulation, acceptance, cognitive flexibility, and interoception) predict or mediate outcomes?
* Non-specific factors: To what extent do treatment expectations and group alliance predict outcomes?

iii. Understanding patients' experience of UP: To explore patients' experience of UP treatment through in-depth qualitative interviews.

Research questions:

* How do participants describe their experience of benefits and challenges with the UP program?
* How do participants describe their experience of change during and after the treatment?

iv.) Understanding transdiagnostic factors in emotional vulnerability and resilience: To explore whether individuals with emotional disorders differ cross-sectionally from healthy controls.

Research question:

- Do patients with emotional disorders differ significantly from healthy controls on measures of emotion regulation, acceptance, cognitive flexibility, and psychophysiological markers (interoception, heart rate variability)?

v.) Examining UP group therapy delivered by novices: To assess whether novice therapists can be trained to deliver UP with high fidelity.

Research question:

- Can novice therapists (i.e., graduate students in clinical psychology under supervision) be trained to high levels of fidelity in delivering the UP group treatment?

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40
* Fulfilling diagnostic criteria for an anxiety disorder and/or unipolar depression (ICD F.3x - 4x)
* Motivated for short-term treatment in group format

Exclusion Criteria:

* Suicidality
* Self-harm
* Severe psychiatric disorder (bipolar disorder, psychosis)
* Substance use disorders
* Use of anxiolytic medication (i.e., benzodiazepines)
* Unstable antidepressant medication (i.e., stable dosage <6 months)
* Other ongoing psychological treatment

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
WHO-5: Wellbeing index | From enrollment to follow-up at 6 months
  The WHO-5 is a self-report measure of positive mental health. It consists of five items that are rated on a 6-point scale from 'All of the time' to 'At no time'. High scores indicate a more positive rating of wellbeing

SECONDARY OUTCOMES:
Work and Social Adjustment Scale | From enrollment to follow-up at 6 months
  The WSAS is a five-item scale that addresses impairments in work/study, home, social life, private leisure activities, and interpersonal relations. Each item is self-rated on a nine-point Likert scale that ranges from "Not at all" (0) to "Severely impaired" (8).
Patient Health Questionnaire (PHQ-9) | From enrollment to follow-up at 6 months
  The PHQ-9 is a nine-item scale measuring depression severity. Each item is self-rated on a four-point Likert scale that ranges from "Not at all" (0) to "Nearly every day" (3).
Generalized Anxiety Disorder Scale (GAD-7) | From enrollment to follow-up at 6 months
  The GAD-7 is a seven-item scale measuring anxiety severity. Each items is self-rated on a four point Likert scale that ranges from "Not at all" (0) to "Nearly every day" (3).
Multidimensional Emotional Disorders Inventory (MEDI) | From enrollment to follow-up at 6 months
  The MEDI is a 49-item scale measuring nine transdiagnostic factors involved in emotional disorders. Each item is self-rated on a nine point Likert scale that ranges from 0 (Not at all characteristic of me) to 8 (Totally characteristic of me). The dimensions measured are Neurotic temperament, positive temperament, depressive mood, autonomic arousal, somatic anxiety, intrusive thoughts, traumatic re-experiencing and avoidance.
Level of Personality Functioning Scale Brief Form (LPFS-BF) | From enrollment to follow-up at 6 months
  The LPFS-BF is a 12-item scale measuring the level of personality functioning based on the Criterion "A" of the alternative model for personality disorders in the DSM-5; Identity, self-direction, empathy and intimacy. Each item is self-rated on a 4-point Likert scale that ranges from 0 (Little or no impairment) to 3 (Severe impairment).
Difficulty in Emotion Regulation Scale (DERS-16) | From enrollment to follow-up at 6 months
  The DERS is a 16-item scale measuring individuals' typical levels of difficulties in emotion regulation. Each item is self-rated on a 5-point Likert scale that ranges from 1 (Almost never) to 5 (Almost always).
Acceptance and Action Questionnaire- version 2 (AAQ-II) | From enrollment to follow-up at 6 months
  The AAQ-II is a 7-item scale measuring experiential avoidance and psychological inflexibility. Each item is self-rated on a 7-point Likert scale that ranges from 1 (Never right) to 5 (Always right). The total score ranges between 0-49. Higher scores indicate less psychological flexibility and more experiential avoidance.
Five Facet Mindfulness Questionnaire (FFMQ) | From enrollment to follow-up at 6 months
  The FFMQ is a 15-item scale measuring mindfulness with regard to thoughts, experiences, and actions in daily life. Each item is self-rated on a 5-point Likert scale that ranges from 1 (Never or rarely true) to 5 (Very often or always true).
Unified Protocol Cognitive Skills Questionnaire (UP-CSQ) | From enrollment to follow-up at 6 months
  The UP-CSQ is a 7-item scale measuring the cognitive skills taught in the UP. Each item is self-rated on a 5-point Likert scale that ranges from 1 (Never) to 5 (Always or when needed)
Multidimensional Assessment of Interoceptive Awareness-2 (MAIA) | From enrollment to follow-up at 6 months
  The MAIA is a 37-item scale measuring interoceptive awareness. Each item is self-rated on a 6-point Likert scale that ranges from 0 (Never) to 5 (Always).
Overall Anxiety Severity and Impairment Scale (OASIS) | At each treatment session through the 12 weeks of treatment
  The OASIS is a 5-item scale measuring the frequency and severity of anxiety, avoidance, work/school/home interference, and social interference due to anxiety. Each item is self-rated on a 5-point Likert scale that ranges from 0 (None, never) to 4 (Extreme, constant). The OASIS is used as an in-session UP measures to examine processes of change
Overall Depression Severity and Impairment Scale (ODSIS) | At each treatment session through the 12 weeks of treatment
  The ODSIS is a 5-item scale measuring the frequency and severity of depression symptoms, avoidance, work/school/home interference, and social interference due to depression. Each item is self-rated on a 5-point Likert scale that ranges from 0 (None/never) to 4 (Extreme/constant). The ODSIS is used as an in-session UP measures to examine processes of change
Unified Protocol Skill Use Scale (UPSUS) | At each treatment session through the 12 weeks of treatment
  The UPSUS is a 7-item scale measuring the frequency with which individuals use UP-skills in distressing situations. Each item is self-rated on a 6-point Likert scale that ranges from 0 (Not at all) to 5 (Nearly all the time). Each item was written to describe core skills taught in each of the five core UP-modules. The UPSUS is used as an in-session UP measure to examine processes of change
Dimension of Skillfulness and Use Scale (DSUS) | At each treatment session through the 12 weeks of treatment
  The DSUS is a 4-item scale measuring the understanding of UP skills learned in the prior session, frequency of skill use, quality of skill use, and effectiveness and skill use. Each item is self-rated on a 5-point Likert scale that ranges from 0 (Not at all) to 4 (Extremely well/every day). The DSUS is used as an in-session UP measures to examine processes of change
Client Satisfaction Questionnaire (CSQ-8) | At final treatment session (week 12)
  The CSQ-8 is an 8-item scale measuring clients' satisfaction with treatment. Each item is scored on a 4-point Likert scale that ranges from 0 to 3.
The Negative Effects Questionnaire (NEQ) | At final treatment session (week 12)
  The NEQ is a 32-item scale measuring adverse or unwanted events during treatment. Each item is designed to assess adverse effects related to psychological treatments. Items are scored on a five-point Likert scale (0-4) and differentiates between treatment-related negative effects and those from external factors.
The Heartbeat Counting Task (HBC) | From enrollment to follow-up at 6 months
  The HBC task evaluates three dimensions of interoception: 1) Interoceptive accuracy in the form of ratio of detected to actual heartbeats, 2) Interoceptive sensibility in the form of self-reported interoception through interviews and questionnaires, and 3) Interoceptive awareness in the form of metacognitive awareness of accuracy, measured by the correlation between confidence and actual performance using receiver operating characteristics (ROC) curve analysis.
Heart Rate Variability (HRV) via a 24-hour ECG Monitoring. | From enrollment to follow-up at 6 months
  24-hour ECG data will be collected using BioPoint sensors from SiFi Labs, which are wearable, small and designed for continuous monitoring. The sensor is placed below the sternum. The data are not intended for clinical evaluation of heart function but suitable for investigating potential changes in HRV before and after psychotherapy in addition to possible differences in HRV in groups of patients with emotional disorders compared to healthy controls.

OTHER OUTCOMES:
Credibility Rating Scale | This scale will be administered only at pre-treatment as a possible predictor of change.
  The version of the Credibility Rating Scale used in this study is a 5-item adapted version of the original Credibility Rating Scale developed by Devilly & Borkovec.
Group Session Rating Scale (GSRS) | At each treatment session through the 12 weeks of treatment
  The GSRS is a 4-item scale measuring each participant's experience of alliance in the UP group therapy. Each item is scored on a visual analog scale, covering the patient's experience of the quality of the relations to both the therapist and the other patients in the group, the personal relevance of the goals and themes of the group session, the fit of the approach utilized in the treatment, and the general experience of being part of the group.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Vøllestad, Ph.D., Principal Investigator — University of Bergen
Locations (1):
- Department of Clinical Psychology, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: No